CLINICAL TRIAL: NCT02302209
Title: Effects of Oxytocin on Familial Interactions
Brief Title: Dyad Oxytocin Study (DOS)
Acronym: DOS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Joshua Woolley, Assistant Professor in Residence, University of California, San Francisco
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 10-04286
Record Dates: First submitted 2014-11-24; First posted 2014-11-26 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Schizophrenia; Autism Spectrum Disorder
Keywords: oxytocin; schizophrenia; autism spectrum disorder
MeSH Terms: conditions — Schizophrenia; Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Oxytocin (Experimental): 40 IU Oxytocin Intranasal
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Saline Nasal Spray
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Drug: Oxytocin
  Other Names: Syntocin
  Arms: Oxytocin
Other: Placebo Comparator
  Arms: Placebo

SUMMARY:
The purpose of the investigators proposed study is twofold: 1) To investigate the role of the affiliative neuropeptide oxytocin in unhealthy interactions in families of patients with schizophrenia and families of patients with autism spectrum disorder, and 2) to investigate whether manipulation of this oxytocinergic system positively influences these family interactions.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for caregiver of patients with schizophrenia, patients with autism spectrum disorder, and healthy controls:
* Age between 18 and 75 years old
* Must have at least 4 hours of contact with the patient per week and be considered a "significant caregiver" by the patient

Inclusion criteria for patients with schizophrenia:

* Between the ages of 14 and 45.
* Patients must have a diagnosis of schizophrenia, schizophreniform disorder, schizoaffective disorder or psychosis- Not Otherwise Specified (NOS).
* Patients must be clinically stable
* No or minor changes to medications in the past week
* Patients must have a primary caregiver
* Inclusion criteria for healthy control child:
* Between the ages of 14 and 45
* Healthy control must have a primary caregiver
* Inclusion criteria for patients with autism spectrum disorder
* Between the ages of 14 and 45
* Patient must have a primary caregiver
* Patients must have a diagnosis of an autism spectrum disorder (ASD) (autism or Asperger's disorder), pervasive developmental disorder (PDD) or pervasive developmental disorder - not otherwise specified (PDD-NOS).

Exclusion Criteria:

Exclusion criteria for all caregivers:

* Female caregivers that state that they are pregnant or have a positive urine pregnancy test
* Caregivers who have significant nasal pathology, atrophic rhinitis, recurrent nose bleeds, or history of cranial-surgical procedures (hypophysectomy)
* Caregivers with significant psychiatric, neurologic, or medical illness
* Exclusion criteria for healthy controls:
* Healthy controls with history of psychiatric or neurological illness
* Exclusion criteria for patients with an autism spectrum disorder:
* Patients with an Intelligence Quotient (IQ) lower than 75
* Exclusion criteria for patients with schizophrenia
* Patients with severe brain trauma

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2011-04; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Negative Expressed Emotion | Continuously for 4 hours after drug adimistration
  We will measure the number of times caregivers show parental criticism, hostility, lack of warmth and emotional over-involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Josh D Woolley, MD/PhD, Principal Investigator — UC San Francisco and SFVAMC
Locations (1):
- University of California, San Francisco, San Francisco, California, United States